CLINICAL TRIAL: NCT02425449
Title: Characterizing Fade Upon Train-of Four Stimulation During Onset and Offset of Neuromuscular Block Produced by Succinlycholine
Brief Title: Fade Upon TOF Stimulation Induced by Succinylcholine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Shashi Bhatt, MD, Associate Professor, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UTIRB 200538
Record Dates: First submitted 2015-04-14; First posted 2015-04-24 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Muscle Relaxants
Keywords: succinylcholine; depolarizing muscle relaxants; pharmacologic effects
MeSH Terms: conditions — Muscle Hypotonia | interventions — Succinylcholine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 01 mg/kg (Experimental): Succinylcholine 0.1 mg/kg will be administered and TOF ratio measured before and after the administration until stable
  Interventions: Drug: Succinylcholine
- 0.15 mg/kg (Experimental): Succinylcholine 0.15 mg/kg will be administered and TOF ratio measured before and after the administration until stable
  Interventions: Drug: Succinylcholine
- 0.2 mg/kg (Experimental): Succinylcholine 0.2 mg/kg will be administered and TOF ratio measured before and after the administration until stable
  Interventions: Drug: Succinylcholine
- 0.25 mg/kg (Experimental): Succinylcholine 0.25 mg/kg will be administered and TOF ratio measured before and after the administration until stable
  Interventions: Drug: Succinylcholine
- 0.3 mg/kg (Experimental): Succinylcholine 0.3 mg/kg will be administered and TOF ratio measured before and after the administration until stable
  Interventions: Drug: Succinylcholine

INTERVENTIONS:
Drug: Succinylcholine — will be administered succinylcholine in a dose of 0.1 mg/kg in Arm 1, 0.15 mg/kg in Arm 2, 0.2 mg/kg in Arm 3, 0.25 mg/kgin Arm 4, 0.3 mg/kg in Arm 5.

SUMMARY:
Muscle relaxants are medications used during surgery to facilitate surgical access. The effect of the muscle relaxant medications is measured by stimulation a motor nerve and measuring the force of the resultant muscle contraction. Based on the mechanism of action, two kinds of muscle relaxants are described. First a nondepolarizing muscle relaxant and the second kind is the depolarizing muscle relaxant. These two kinds of muscle relaxants can be distinguished by rapidly stimulating the nerve 4 times over 2 seconds (Train of four or TOF). The nondepolarizing muscle relaxants produce fade ie successive muscle contractions are less forceful than the preceding ones. Whereas the depolarizing muscle relaxants are generally believed to produce four contractions of equal strength. However, there is some indication that this may not be entirely correct. There is evidence that depolarizing muscle relaxants also may produce fade. The investigators are conducting the following study to determine if indeed depolarizing muscle relaxants produce fade. The investigators would also like to characterize the fade ie differences during onset and offset of the block and the effect of the dose on the degree on the fade.

DETAILED DESCRIPTION:
Muscle relaxants are frequently employed during anesthesia. These medications may be employed to facilitate tracheal intubation, mechanical ventilation or to allow better surgical access. All muscle relaxants act at the neuromuscular junction. Based on the mechanism of action, two kinds of muscle relaxants have been defined1. Nondepolarizing muscle relaxants are competitive antagonists of the neurotransmitter acetylcholine (Ach) at the neuromuscular junction. The second kind of muscle relaxant is the depolarizing muscle relaxant and succinylcholine is the only muscle relaxant in this class that is clinically used. The mechanism of action of succinylcholine is less clear. Succinylcholine appears to mimic the actions of acetylcholine but results in a longer duration of depolarization of the post synaptic membrane1.

The degree of muscle relaxation produced by these muscle relaxants is measured by stimulating a motor nerve and measuring either the force of the muscle contraction produced or its compound muscle action potential (CMAP). As the muscle relaxation increases, the force of muscle contraction or the amplitude of the electromyogram (EMG) is correspondingly reduced.

On occasion, to measure the degree of muscle weakness or paralysis caused by a muscle relaxant, instead of a single stimulus, trains of stimuli are applied2. One method of repetitive stimulation is to apply four stimuli over a two second period. This method of nerve stimulation is called Train-of-Four (TOF). When this form nerve stimulation (TOF) is applied to patients who have been given nondepolarizing muscle relaxants -there is fade. Fade means that the force of successive muscle contractions is less than the preceding contraction3. The second contraction is less than the first, the third less than the second and so on. The degree of fade appears to have some reasonably well defined relationship to the degree of relaxation produced3.

The classic teaching in the anesthetic literature is that depolarizing muscle relaxants do not produce fade upon repetitive stimulation. It means that upon repetitive stimulation, the successive contractions are similar. This is one of the defining features of a depolarizing block and is called a Phase I block. The traditional teaching is that when a depolarizing muscle relaxant is administered in large or repetitive doses, a Phase II block develops. The phase II block has characteristics similar to those of a nondepolarizing muscle relaxant (ie fade on repetitive or TOF stimulation). De Jong and Freund first proposed that this differentiation between deplolarizing and nondepolarizing block based upon fade may not be as clear cut. These investigators demonstrated that succinylcholine caused fade upon repetitive stimulation right from the outset of the neuromuscular block. Other investigators have also demonstrated that succinylcholine causes fade from the initiation of the neuromuscular block. If it can be conclusively demonstrated that succinylcholine causes fade, then fade would be less useful in differentiating a depolarizing from a nondepolarizing block. We have previously investigated and defined the fade caused by nondepolarizing muscle relaxants. Using the experience we have gained in studying fade with nondepolarizing muscle relaxants, we would like to now define the characteristics of fade (if any) caused by succinylcholine.

Method: We intend to enroll fifty healthy adults, 18-60 years of age of either sex who are scheduled to undergo a surgical procedure under general anesthesia. Only subjects with a BMI <25 Kg/m2 will be enrolled. Only subjects free from any hepatic or renal disease will be included. We will exclude any subjects with known allergy to succinylcholine, family history of malignant hyperthermia or any history of skeletal myopathy. We will also exclude subjects that have recently sustained burns, or any illness resulting denervation injury (paraplegia or hemiplegia).

The subjects will give an informed consent prior to the participation in the study. All patients will receive 2 mg of midazolam for premedication. Anesthesia will be induced with the intravenous administration of fentanyl 5-6 µg/kg and propofol 2-3 mg/kg. Following tracheal intubation, anesthesia will be maintained with 70% nitrous oxide in oxygen supplemented with an infusion of propofol (120 -150 µg/kg/min). Ventilation will be controlled to maintain normocapnia (end-tidal carbon di oxide 35-40 mmHg).

After the commencement of the anesthesia monitoring of neuromuscular transmission will be commenced. Ulnar nerve at the wrist will be stimulated in a TOF sequence (2 Hz every 12 seconds). The resultant force of contraction of the adductor pollicis will be recorded using a mechanomyograph. After obtaining a stable muscle contraction, succinylcholine will be administered. The subjects will be randomly allocated to one of five groups. Group 1 will receive 0.1 mg/kg, group 2 -0.15 mg/kg, group 3 -0.2 mg/kg, group 4 -0.25 mg/kg, group 5 -0.3 mg/kg. Muscle contraction will be recorded until the force of muscle contraction returns to baseline (6-8 minutes). At this time the study will be concluded. Further conduct of the anesthetic will be at the discretion of the subject's primary anesthesiologist.

Data Analysis: We intend to plot the force of all four muscle contractions from immediately preceding the injection succinylcholine to complete recovery of the muscle contraction. We would then plot the force of the first twitch (T1) against the ratio of the fourth to the first twitch (T4/T1 ratio) for each individual subject. This plot will allow us to determine if there is any difference in fade characteristics between onset and offset of muscle relaxant effect.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS I or II,
* 18-60 years of age of either sex,
* with a BMI<25Kg/m2

Exclusion Criteria:

* presence of any disease involving the neuromuscular system.
* Presence of any neurologic illness eg . Paraplegia or hemiplegia, spinal cord injuries, stroke, multiple sclerosis.
* No liver or kidney disease.
* Known allergy to succinylcholine.
* Family history of malignant hyperthermia.
* Known pseudocholinesterase deficiency.
* Any skin burns within the last 1 year.

We would also exclude subjects with;

* Central core disease,
* duchenne or Becker muscular dystrophy,
* osteogenesis imperfecta,
* Noonan syndrome,
* arthrogryposis multiplex,
* congenital,
* myotonia,
* neuroleptic malignant syndrome,
* multiminicore disease,
* King Denborough syndrome,
* Native American myopathy,
* hypokalemic periodic paralysis or
* a history of rhabdomyolysis.

We would also exclude any subject with a history of cardiac arrhythmias.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shashi Bhatt, MD, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: 0.1 mg/kg of succinylcholine arm
  Succinylcholine: will be administered succinylcholine in a dose of 0.1 mg/kg in Arm 1, 0.15 mg/kg in Arm 2, 0.2 mg/kg in Arm 3, 0.25 mg/kgin Arm 4, 0.3 mg/kg in Arm 5.
- Arm 2: 0.15 mg/kg of succinycholine arm
  Succinylcholine: will be administered succinylcholine in a dose of 0.1 mg/kg in Arm 1, 0.15 mg/kg in Arm 2, 0.2 mg/kg in Arm 3, 0.25 mg/kgin Arm 4, 0.3 mg/kg in Arm 5.
- Arm 3: 0.2 mg/kg of succinylcholne arm
  Succinylcholine: will be administered succinylcholine in a dose of 0.1 mg/kg in Arm 1, 0.15 mg/kg in Arm 2, 0.2 mg/kg in Arm 3, 0.25 mg/kgin Arm 4, 0.3 mg/kg in Arm 5.
- Arm 4: 0.25 mg/kg succinylcholine arm
  Succinylcholine: will be administered succinylcholine in a dose of 0.1 mg/kg in Arm 1, 0.15 mg/kg in Arm 2, 0.2 mg/kg in Arm 3, 0.25 mg/kgin Arm 4, 0.3 mg/kg in Arm 5.
- Arm 5: 0.3 mg/kg succinylcholine arm
  Succinylcholine: will be administered succinylcholine in a dose of 0.1 mg/kg in Arm 1, 0.15 mg/kg in Arm 2, 0.2 mg/kg in Arm 3, 0.25 mg/kgin Arm 4, 0.3 mg/kg in Arm 5.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5
Started | 0 | 4 | 5 | 5 | 5
Completed | 0 | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Total
Number analyzed (Participants) | 0 | 4 | 5 | 5 | 5 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 35.3 (6.7) | 38.4 (11.1) | 37.4 (6.2) | 36.2 (12.8) | 36.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 3 | 3 | 4 | 11
  Male |  | 3 | 2 | 2 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Fade on Train of Four Stimulation
Description: We stimulated the ulnar nerve at the wrist four times (over 1.5 seconds) every 20 seconds. We measured the ratio of the fourth contraction to the first contraction before and after the administration of succinylcholine. Before administering succinylcholine the ratio is normally one. After the administration of succinylcholine the first contraction diminishes, but the fourth contraction diminishes even more. This results in a ratio of T4 to T1 being less than one. The lowest ratio recorded after the administration after the administration of succinylcholine is reported as our outcome measure.
Time Frame: for the duration of the effect of succinylcholine generally expected to be 6-10 minutes
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5
Number analyzed (Participants) | 0 | 4 | 5 | 5 | 5
Ratio |  | 0.85 (0.02) | 0.64 (0.04) | 0.66 (0.09) | 0.68 (0.04)

ADVERSE EVENTS:
Time Frame: Adverse event were collected for the duration of the surgical procedure generally 1- 2 hours.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/4 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/4 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/0 | 0/4 | 0/5 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes